CLINICAL TRIAL: NCT05323071
Title: Comparison of the Effectiveness of Administering 24% Oral Sucrose Two Minutes Before Versus at the Same Time in the Performance of a Painful Procedure in the Neonate.
Brief Title: Comparison of the Efficacy of Oral Sucrose Administration at Two Different Times of a Painful Procedure in Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oihana Lopez Alonso (Network)
Responsible Party: Sponsor-Investigator, Oihana Lopez Alonso, Neonatal unit nurse, Bioaraba Health Research Institute
Organization: Bioaraba Health Research Institute (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Expte. 2021-025
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Sucrose will be administered 2 minutes before the puncture following the current protocol of the unit. Venous or arterial puncture will be performed only in case it is required for therapeutic or care purposes.
  Interventions: Other: Sucrose 24%
- Experimental Group (Experimental): The administration of the sucrose dose is started by means of a syringe. Once 50% of the dose has been administered, puncture will be performed. The remaining 50% will be administered during the puncture. The pacifier will be left in the mouth until the end of the procedure, facilitating the non-nutritive sucking of the neonate.
  Interventions: Other: Sucrose 24%

INTERVENTIONS:
Other: Sucrose 24% — According to the age of the newborn:
  24-26 weeks : 0.1 mL, 27-31weeks : 0.25 mL, 32-36 weeks : 0.5 mL, >37 weeks : 1 mL

SUMMARY:
The objective of this study is to compare the use of 24% sucrose in pain control in neonates from 32 weeks of gestation onwards according to the time of administration of sucrose in venous and arterial puncture for blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Neonates whose parents and/or guardians have signed the informed consent form.

Exclusion Criteria:

* Neonates connected to invasive mechanical ventilation.
* Neonates presenting any type of neurological alteration or showing signs of irritability prior to the puncture.
* Neonates who have received sedation.
* Neonates presenting withdrawal syndrome.

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Pain during a painful procedure | 15 seconds after extraction
  The primary variable is pain, and will be measured by the Premature Infant Pain Profile-Revised (PIPP-R) scale. The score ranges from 0 (no pain or minimal pain) to 21 (maximum pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Araba-Sede Txagorritxu, Vitoria-Gasteiz, Alava, Spain